CLINICAL TRIAL: NCT03317236
Title: Bioequivalence Study of Quetiapine in Healthy Volunteers, After Administering a Single Dose of the Test Extended Release Formulation, Kemoter XR With Respect to the Reference Product, Etiasel XR ® From AstraZeneca S.A.
Brief Title: Bioequivalence Study of Two Extended Release Formulations Containing 50 mg of Quetiapine.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratorio Elea Phoenix S.A. (Industry)
Collaborators: DominguezLab S.R.L. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PRO-BEQ-QTP-002-V.01
Record Dates: First submitted 2017-10-18; First posted 2017-10-23 (Actual); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: Healthy
Keywords: Bioequivalence; Quetiapine
MeSH Terms: interventions — Quetiapine Fumarate

STUDY DESIGN:
Intervention Model Description: Single-dose, two-way crossover.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reference - Test (Experimental): A new extended release formulation containing quetiapine 50 mg (T) followed by a branded formulation (R).
  Interventions: Drug: Quetiapine
- Test - Reference (Experimental): A branded formulation (R) followed by a new extended release formulation containing quetiapine 50 mg (T).
  Interventions: Drug: Quetiapine

INTERVENTIONS:
Drug: Quetiapine — A fixed 50 mg exteded release formulation.

SUMMARY:
Bioequivalence study of quetiapine in healthy volunteers, comparing the test extended release formulation, Kemoter XR with respect to the reference product, Etiasel XR ® from AstraZeneca S.A., under a single-dose, two-way crossover design.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Healthy volunteers according to medical history, physical exam, clinical laboratory, chest X-rays and ECG.
* Gender: males and non pregnant females
* Age: 18 to 55 years.
* Body mass index: 19 to 27 kg/m^2.

Exclusion Criteria:

* History of liver or renal disease, or psychiatric disorders.
* History of drug or alcohol abuse during the previous two years.
* Smokers of more than 10 cigarrettes a day.
* Any kind of medicines taken during the previous two weeks.
* Any history of disease or disorders clinically significant according to the Principal Investigator.
* Abnormal ECG.
* Abnormal chest X-ray.
* Hypersensitivity to quetiapine or excipients within the formulations.
* Positive diagnostic test for HIV or hepatitis A, B or C virus.
* Breast feeding females.
* Positive beta-HCG test.
* Positive drug test in urine.
* Participation in clinical trials in the previous three months.
* Blood donation in the previous three months.
* Clinically significant laboratory results.
* Subjects seeking to initiate any medical or pharmacological treatment.
* Subjects unwilling to keep fasting or diet indications.
* Uncooperative subjects.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Cmax | 36 hours
  Maximum plasma concentration
AUC | 36 hours
  Area under curve

CONTACTS AND LOCATIONS:
Overall Officials: María C Fritz, MD, Principal Investigator — DominguezLab S.R.L.
Locations (1):
- DominguezLab, Paraná, Entre Ríos Province, Argentina

IPD SHARING:
Plan to Share IPD: No